CLINICAL TRIAL: NCT06668636
Title: Examining the Effectiveness and Implementation of the Emergency Department Patient-Activated Transition to Care At Home (ED-PATCH) Tool: a Mixed Methods Hybrid Type 1 Design Study
Brief Title: Examining the Effectiveness and Implementation of the Emergency Department Patient-Activated Transition to Care At Home Tool
Acronym: ED-PATCH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Janet Curran, Quality and Patient Safety Research Chair, IWK Health Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IWK-REB-1030763; 190304 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Emergency Department Discharge Communication
Keywords: emergency department; discharge communication; discharge instructions; mobile applications
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: This study will employ an interrupted time series design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-Implementation (No Intervention): This arm of the study will occur before ED-PATCH has been implemented. Patients will receive usual discharge communication.
- Post-Implementation (Experimental): This arm of the study will occur after ED-PATCH has been implemented.
  Interventions: Behavioral: ED-PATCH

INTERVENTIONS:
Behavioral: ED-PATCH — Participants will access ED-PATCH using their personal mobile device and use it to track important information throughout their visit. The summary will be checked by a healthcare provider and corrected, if necessary, before being locked and sent to the patient or caregiver to keep for their own records.
  Arms: Post-Implementation

SUMMARY:
The goal of this clinical trial is to examine the effectiveness and implementation of the Emergency Department Patient-Activated Transition to Care at Home (ED-PATCH) tool, which is used by patients to manage information during their visit to the emergency department. The main aims of the trial are:

* To study whether ED-PATCH works well in Canadian emergency department settings
* To understand the context and strategies impacting the implementation of ED-PATCH in Canadian emergency department settings

ED-PATCH is an electronic tool accessed using a smartphone or tablet that patients and caregivers can use to create their own summary of what happened during their visit to the emergency department. Using a questionnaire format, the tool prompts users to enter information about their symptoms, tests and procedures done during the visit, diagnosis, medications given, and their plans after leaving the emergency department. A healthcare provider checks that the information is correct before the summary is locked and emailed to the patient.

Researchers will compare data collected before ED-PATCH is launched and after it is launched to learn if the tool reduces return visits to the emergency department and other outcomes such as participants' stress, memory and understanding of their visit, health status, and care experiences.

DETAILED DESCRIPTION:
When patients and caregivers leave the emergency department (ED) without fully understanding the care provided and the information shared during their visit, it can impede their ability to effectively manage their care at home. Effective discharge communication can reduce return visits, helping keep ED patient volumes manageable, and improve patient and caregiver outcomes. Opportunities exist to improve patient-provider discharge communication and ensure patients and caregivers have mastery of the knowledge needed to manage their health condition after they leave the ED. Novel health technology solutions have shown some potential to enhance discharge communication practice.

Emergency Department Patient-Activated Transition to Care at Home (ED-PATCH) is a discharge communication tool that is activated and managed by patients or their caregivers to record important information shared during the ED visit. Patients receive ED-PATCH in the waiting room or immediately upon placement in the assessment room and use it to track important information throughout their visit. The tool will support tracking information shared during the ED visit including (1) information about diagnosis; (2) details about treatments, tests and procedures; (3) reconciled and new medications; and (4) treatment plans including expected course of illness, signs and symptoms to watch for and when to return to the ED. Prior to discharge, the patient or caregiver shares the summary of their notes with an ED provider who confirms or clarifies the information captured. The patient-generated discharge summary is then sent electronically to the patient or caregiver to be added to their own personal health record.

The primary aim of this study is to evaluate the effectiveness of ED-PATCH in Canadian adult and pediatric emergency department settings. The secondary aim is to better understand the context and strategies for implementation of ED-PATCH in Canadian adult and pediatric emergency department settings. The objectives are to (1) evaluate the effectiveness of ED-PATCH on patient recall and comprehension of information during an emergency department visit; (2) evaluate the effectiveness of ED-PATCH on patient experience with emergency care; (3) evaluate the impact of ED-PATCH on health care provider and health system outcomes; (4) explore the determinants (patient/caregiver, provider, and system factors) of ED-PATCH adoption in emergency practice settings; and (5) describe the implementation strategies employed to promote uptake of ED-PATCH.

Effectiveness and implementation will be investigated concurrently in this study using a mixed methods hybrid type 1 effectiveness-implementation design with an integrated knowledge translation (iKT) approach. Effectiveness-implementation hybrid designs have a dual focus on clinical effectiveness and implementation. Quantitative measures (e.g., rate of ED admissions) will be used to evaluate intervention effectiveness while mixed methods (qualitative and quantitative) will be used to describe barriers and enablers to implementation and/or evaluate implementation outcomes such as feasibility, reach, adoption, and sustainability.

The investigators will use an interrupted time series (ITS) design to address the first two objectives and estimate the effect of ED-PATCH on the aggregate primary outcome measures at ED sites in Nova Scotia, Quebec, Alberta, and Ontario. Primary and secondary outcomes will be measured up to 18 months pre-implementation and 18 months post-implementation. The investigators will address the remaining objectives by tracking implementation of ED-PATCH and conducting semi-structured, qualitative interviews with a subset of participants and ED providers.

Integration of effectiveness and implementation findings will be guided by RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance), a systems-level evaluation framework used extensively to assess intervention implementation and sustainability. RE-AIM will be adapted using a health equity lens to strengthen the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Youth and adults aged 14 years and older are eligible to participate on their own behalf; caregivers or support people aged 14 years and older are eligible to participate on behalf of children younger than 14 years old
* Seeking emergency care at participating sites on their own behalf or as a caregiver or support person for another patient
* Discharged home from the ED
* Able to understand and read English or French
* Meet Canadian Triage Acuity Scale (CTAS) between 2-5
* Provide informed consent

Exclusion Criteria:

* Infants and children aged under 14 years are not eligible to participate on their own behalf
* Admitted to hospital after seeking emergency care
* Unable to understand or read English or French
* CTAS of 1
* Not providing informed consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Monthly Rate of ED and Hospital Readmissions | 7 days post-index visit
  Monthly rate of emergency department and hospital readmissions (composite) at 7 days post-index visit, per every 100 visits, assessed of all available visits at each site.

SECONDARY OUTCOMES:
Patient-Reported Outcomes (PROM-ED) | At baseline and 72 hours after discharge
  The PROM-ED questionnaire will be used to measure patient-centered outcomes of importance during transitions in emergency care across four domains: symptom relief, understanding of their health concern, reassurance, and having a plan they can follow.
Perceived Stress | At baseline
  Patients' perceived stress will be measured during the ED visit using the visual analogue scale (VAS) for stress, with which participants rate their stress level on a scale from 0 (no stress) to 10 (worst possible stress).
Patient Experiences of Care Transitions (ED CAHPS) | 72 hours after discharge
  Patient experiences of care transitions will be measured using the Emergency Department Consumer Assessment of Healthcare Providers and Systems (ED CAHPS) survey which includes 35 questions that focus on communication and coordination of care during the visit.
Recall and Comprehension Survey of Information Shared During the ED Visit | 72 hours and 7 days after discharge
  A survey created for the study will measure patient or caregiver's recall and comprehension of four key areas related to their care: 1. Diagnosis; 2. Procedures and diagnostic tests undertaken during the index visit; 3. Medication administered during their visit and medication prescribed on discharge; and 4. Details regarding follow-up. The survey responses will be corroborated with details about the ED visit from the patient chart.
Health Care Utilization (Length of Stay, Return Visits, Hospital Admissions) | 72 hours after discharge, 7 days after discharge, 30 days after discharge
  Hospital administrative databases will be used to calculate length of stay (total time from assessment in triage to discharge), ED return visits within 72 hours, ED return visits at 7 days, ED return visits at 30 days, and hospital admissions at 7 days.
Implementation Tracking | 18 months post-implementation
  The Framework for Reporting Adaptations and Modifications-Enhanced Implementation Strategy (FRAME-IS) will guide tracking the nature of any modifications and adaptations to the implementation strategy, when they occurred, who participated in the decision to modify, and the reasons why the changes were made.
Patient and Provider Perceptions of Implementation | Patient participants: 4 weeks post-discharge; Provider participants: 8 weeks after ITS closure
  A semi-structured qualitative interview guide will be used to solicit patient and provider perspectives on how ED-PATCH was implemented.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - IWK Health, Halifax, Nova Scotia
  - Valley Regional Hospital, Kentville, Nova Scotia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified datasets generated during the proposed study may be made available on request to those with a methodologically sound proposal and pending ethics approval.
Supporting Information: Study Protocol, ICF
Time Frame: 2028 (planned)
Access Criteria: Those with a methodologically sound proposal and ethics approval can contact the Principal Investigators to request the IPD.